CLINICAL TRIAL: NCT01263834
Title: The Results of Adjunctive Intraoperative Bevacizumab Injection on Trabeculectomy Outcome: A Randomized Controlled Trial
Brief Title: Results of Adjunctive Intraoperative Bevacizumab Injection on Trabeculectomy Outcome
Acronym: Bevacizumab
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Weerawat Kiddee, Dr.Weerawat Kiddee, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC 53-296-02-1-2
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Glaucoma
Keywords: Trabeculectomy; bevacizumab; intraocular pressure
MeSH Terms: conditions — Glaucoma | interventions — Bevacizumab; Mitomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mitomycin c (Active Comparator): Mitomycin C soaked cellulose dose 0.4 mg/ml with 3 minutes of application
  Interventions: Drug: Mitomycin C
- Bevacizumab (Experimental): Bevacizumab injection of 1.25m/0.05 cc + Mitomycin C soaked cellulose dose 0.4 mg/ml with 3 minutes of application
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab injection of 1.25m/0.05 cc + Mitomycin C soaked cellulose dose 0.4 mg/ml with 3 minutes of application
  Other Names: Avastin
  Arms: Bevacizumab
Drug: Mitomycin C — Mitomycin C soaked cellulose dose 0.4 mg/ml with 3 minutes of application
  Other Names: MMC
  Arms: Mitomycin c

SUMMARY:
The purpose of this study is to evaluate the adjunctive effect of intratenon Bevacizumab on the result of trabeculectomy in primary term of intraocular pressure (IOP).

DETAILED DESCRIPTION:
Prospective interventional clinical trial

Single center, outcome assessor-masked, active control, randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma with primary mmc-trabeculectomy indication

Exclusion Criteria:

* combined phacoemulsification with trabeculectomy
* no more than 6 month of cataract surgery before trabeculectomy
* revised trabeculectomy
* active uveitic glaucoma
* neovascular glaucoma
* par planar vitrectomy
* conjunctival surgery
* allergy to bevacizumab or mitomycin C
* ischemic heart disease
* cerebrovascular disease
* renal failure
* liver failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | 6 month

SECONDARY OUTCOMES:
Bleb characteristic grading | 6 month
systemic Blood pressure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Weerawat Kiddee, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Glaucoma unit , Department of Ophthalmology Faculty of Medicine Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand